CLINICAL TRIAL: NCT02492659
Title: Clinical Research of Femtosecond Laser-Assisted Cataract Surgery: Randomized Clinical Trial
Brief Title: Clinical Research of Femtosecond Laser-Assisted Cataract Surgery
Acronym: FLACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, A-Yong Yu, clinical professor, Wenzhou Medical University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Femtosecond Laser
Record Dates: First submitted 2015-06-19; First posted 2015-07-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Cataracts
Keywords: femtosecond laser
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- trial group (Experimental): the trial group underwent femtosecond laser-assisted cataract surgery
  Interventions: Procedure: femtosecond laser-assisted cataract surgery
- control group (Other): the control group underwent conventional phacoemulsification
  Interventions: Procedure: conventional phacoemulsification

INTERVENTIONS:
Procedure: femtosecond laser-assisted cataract surgery — the femtosecond laser platform was used to generate capsulotomy with a diameter as described above in the control group, and lens fragmentation into 6 segments.
  Arms: trial group
Procedure: conventional phacoemulsification — continuous curvilinear capsulorhexis was performed with capsulorrhexis forceps. Following hydrodissection, phacoemulsification of the nucleus, aspiration of the residual cortex and capsular polishing were performed using a phacoemulsification machine
  Arms: control group

SUMMARY:
Since femtosecond laser was approved for cataract surgery by FDA in 2010, femtosecond laser assisted cataract surgery (FLACS) has demonstrated high precision of capsulotomy, reduced phacoemulsification power and time, and comparable refractive outcome in clinic.

It is still unknown whether there are toxic substances produced due to photochemical or high-energy physical effect of femtosecond laser during FLACS.

DETAILED DESCRIPTION:
Phacoemulsification is one of the main surgical procedures for cataract surgery owing to the advantages of small incisions and rapid recovery. However, the surgical outcome of phacoemulsification can be negatively affected due to the problem of accuracy and repeatability for capsulorhexis, and the corneal endothelial cell damage by ultrasound energy.To overcome those problems from the phacoemulsification, femtosecond laser-assisted cataract surgery (FLACS) had been used in the past few years and showed unique advantages.

The purpose of this study is to investigate the preliminary clinical outcomes of femtosecond laser-assisted cataract surgery.This prospective comparative study enrolled consecutive patients,will be randomly assigned to trial group underwent FLACS and control group underwent conventional cataract surgery.

The phacoemulsification time, energy, and complications during operation were recorded.

The anterior capsule and aqueous humor were collected. Morphology of the cutting edge and cells of anterior capsule was assessed by light microscopy. The proteins in the aqueous humor were identified by mass spectrometry . Electrolyte in the aqueous humor was detected by a chemistry analyzer. Postoperative refraction at 1 day, 1 week, 1 and 3 months, the capsulorhexis size and corneal endothelial density at 1 and 3 months were also measured.

ELIGIBILITY:
Inclusion Criteria:

1. normal cornea
2. dilated pupillary diameter greater than 6mm
3. no local or systemic contraindications to cataract surgery

Exclusion Criteria:

1. corneal pathological changes
2. glaucoma
3. ocular inflammation
4. previous ocular trauma or surgery

Ages: 38 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
the proteins in the aqueous humor after femtosecond laser operation | day 1

SECONDARY OUTCOMES:
the electrolyte in the aqueous humor after femtosecond laser operation | day 1
morphology of the anterior capsule after femtosecond laser operation | day 1

OTHER OUTCOMES:
phacoemulsification energy | in operation
phacoemulsification time | in operation
postoperative refraction | day 1,after one week
the capsulorhexis size | after one month,after three month
corneal endothelial density | after one month,after three month

CONTACTS AND LOCATIONS:
Overall Officials: A-Yong Yu, PhD, Principal Investigator — Wenzhou Medical University
Locations (1):
- Eye Hispital of Wenzhou Medical University, Wenzhou, Zhejiang, China